CLINICAL TRIAL: NCT00662051
Title: Oral Contraceptives and Asthma Control
Status: Withdrawn | Type: Observational
Sponsor: University of Kentucky (Other)
Collaborators: American College of Allergy, Asthma and Immunology (Other)
Responsible Party: Sponsor
Other Study IDs: 07-0589-F6A
Record Dates: First submitted 2008-04-15; First posted 2008-04-21 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Asthma; Regulatory T Cell Function
Keywords: Asthma; Exhaled Nitric Oxide; Asthma Control Test
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- OCP Users
- Non-users of OCPs

SUMMARY:
Asthma is a chronic inflammatory disorder of the airways affecting approximately 15 million individuals in the U.S. The rate of asthma exacerbations among women is twice that of men after adolescence, and a large proportion of females with asthma report worsened asthma symptoms during different phases of the menstrual cycle. Hormonal influences have been hypothesized to account for these differences. Decreased peak flow rates and increased symptoms have been found in females during the premenstrual phase of the menstrual cycle when estrogen and progesterone levels are low. Estrogen and progesterone have both been found to reduce smooth muscle contractility and increase bronchial smooth muscle relaxation. A perimenstrual shift toward a Th2 (allergic) phenotype characterized by a decreased interferon-gamma to interleukin-10 ratio has been demonstrated in healthy women not using oral contraceptives compared to midcycle; however, the effect was blunted in healthy oral contraceptive pill users, implying hormonal modulation of the allergic phenotype. Several case reports have demonstrated a therapeutic benefit of oral contraceptives in decreasing asthma exacerbations and corticosteroid requirements. Human studies have demonstrated that estrogen decreases pro-inflammatory cytokine generation, neutrophil recruitment, and inhibits inducible nitric oxide synthase activity, which could lead to lower exhaled nitric oxide levels.

The measurement of the fractional concentration of exhaled nitric oxide (FENO) is a non-invasive method to assess airway inflammation in adults and children with asthma. The hypotheses of the current study are that women using oral contraceptives will have lower FENO levels and better asthma control as assessed by the Asthma Control TestTM during different phases of the menstrual cycle. This study may identify clinically important changes in FENO levels and asthma control during the menstrual cycle and modification of these effects by oral contraceptive pills. This data may lead to future studies aimed at identifying therapeutic roles for hormones in asthma therapy in women.

ELIGIBILITY:
Inclusion Criteria:

* Asthmatic
* Female
* Aged 18-45
* User of combination oral contraceptive pills OR non-user of any hormonal contraception

Exclusion Criteria:

* Smoker
* Other underlying lung disease (i.e., emphysema, cystic fibrosis, lung cancer)
* User of oral contraceptives that are not combination (estrogen + progesterone) pills
* User of non-oral hormonal contraception
* Have been treated in the prior 4 weeks with oral steroids
* Have had a respiratory infection in the prior 4 weeks
* Asthma under poor control at study entry
* Presence of severe asthma

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects will be recruited from University of Kentucky clincis and the surrounding community.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Exhaled Nitric Oxide Levels | 2 months

SECONDARY OUTCOMES:
Asthma Control Test Scores | 2 months
Regulatory T Cell Activity | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: James Temprano, MD, MHA, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States